CLINICAL TRIAL: NCT04745923
Title: Fear of COVID-19 and Physical Activity Level in Patients with Chronic Kidney Disease During COVID-19 Pandemic
Brief Title: Physical Activity Level in Patients with Chronic Kidney Disease During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Research assistant, Hacettepe University
Other Study IDs: GO 21/127
Record Dates: First submitted 2021-02-06; First posted 2021-02-09 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Chronic Kidney Diseases
Keywords: Fear; Quality of life; Anxiety; Depression
MeSH Terms: conditions — COVID-19; Renal Insufficiency, Chronic; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with chronic kidney disease: Having been diagnosed with chronic kidney disease
- Healthy individuals: Healthy individuals without chronic disease

SUMMARY:
In the literature, there are no studies evaluating fear of COVID-19, anxiety, depression, physical activity, fear of movement and quality of life in patients with chronic kidney disease during COVID-19 pandemic. The investigators will evaluate these parameters in patients with chronic kidney disease and compare the findings of healthy individuals during COVID-19 pandemic

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with chronic kidney disease
* Being clinically stable
* Volunteering to participate in the research

Exclusion Criteria:

* Having a cognitive problem
* Not being literate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy individuals between 18-65 years old, who are diagnosed with chronic kidney disease, and whose local language is Turkish will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fear of COVID-19 | 5 minutes
  COVID-19 phobia will be evaluated using Fear of COVID-19 Scale.
Physical activity | 5 minutes
  Physical activity level will be evaluated using International Physical Activity Questionnaire - Short Form (IPAQ-SF).

SECONDARY OUTCOMES:
Qol | 10 minutes
  Quality of life will be evaluated using SF-36
Anxiety and depression | 5 minutes
  Anxiety and depression will be evaluated using Hospital Anxiety and Depression scale (HADS).
Fear of movement | 10 minutes
  Fear of movement will be evaluated using the Tampa Scale for Kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, MSc, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Tolga Yildirim, MD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)